CLINICAL TRIAL: NCT05744362
Title: Outcome of Transanal Specimen Extraction Surgery for Elderly Colorectal Cancer Patients: a National Database Study in China of 1395 Cases
Brief Title: Outcome of Transanal Specimen Extraction Surgery for Elderly Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Zhang Hao, Clinical Professor, The Second Affiliated Hospital of Harbin Medical University
Other Study IDs: KY2022-313
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: survival
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective analysis of a cohort of elderly CRC patients (aged ≥ 65 years) underwent transanal-NOSES between August 2008 and February 2022 was constructed. Data were obtained from China NOSES Database (CNDB). The primary outcomes included time to first flatus, postoperative hospital stays, 30-day postoperative complication and hospital mortality. The secondary outcomes were overall survival (OS) and disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed as T1-4N0-2M0 colorectal cancer pathologically

patients underwent transanal-NOSES

patients aged 65 years or older

Exclusion Criteria:

patients with multiple primary colorectal cancer

patients with total colectomy

patients without complete data

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: elderly CRC patients with transanal-NOSES surgery
Sampling Method: Probability Sample
Enrollment: 1395 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4-year
  Time of death from any cause after survival

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China